CLINICAL TRIAL: NCT06890858
Title: A Clinical Study on Fasudil Hydrochloride for Treatment of Gene-Specific Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Yang, MD, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024213
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Fasudil Hydrochloride
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fasudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Fasudil Hydrochloride (Experimental): The specific method is as follows: (1) Administer the standard treatment plan combined with intravenous injection of Fasudil 30mg/2-3 times/day to the enrolled ovarian cancer patients, with the same duration of use as the standard treatment plan. (2) Observe the treatment effect of patients after 2-3 treatment cycles, with the main endpoint being the objective response rate (ORR) and the safety of drug use. The secondary endpoint is the PFS time after combined use of fasudil.
  Interventions: Drug: Fasudil Hydrochloride

INTERVENTIONS:
Drug: Fasudil Hydrochloride — Exploring whether the study of using Exploring whether the study of using Fasudil Hydrochloride for the treatment of gene specific ovarian cancer can be used to predict the sensitivity of immunotherapy for non-small cell lung cancer and other tumors for the treatment of gene specific ovarian cancer can be used to predict the sensitivity of immunotherapy for non-small cell lung cancer and other tumors

SUMMARY:
This is a prospective study investigating whether the research on Fasudil Hydrochloride in the treatment of gene-specific ovarian cancer can be applied to predict sensitivity to immunotherapy in non-small cell lung cancer (NSCLC) and other tumors. The study plans to enroll 20 patients with A/A genotype ovarian cancer for treatment evaluation.

DETAILED DESCRIPTION:
Ovarian cancer is a common gynecological malignancy with the highest mortality rate among gynecological cancers. The poor prognosis and low survival rate in advanced-stage patients primarily contribute to its high mortality. Current clinical management of malignant ovarian tumors relies on postoperative chemotherapy and radiotherapy, which impose significant harm to the human body and offer limited improvement in patient prognosis. Additionally, the diagnostic and therapeutic cycle for malignant ovarian cancer is prolonged and unpredictable, predominantly focusing on post-surgical interventions.

In our preliminary studies, we identified that the A allele of SNP-rs1192691, associated with ovarian cancer prognosis, promotes ovarian cancer cell proliferation and invasion by activating the Rho signaling pathway. The Rho signaling pathway inhibitor Fasudil has been shown to effectively suppress the proliferation and invasion of A/A genotype tumor cells in murine models. This study aims to investigate the therapeutic efficacy of Fasudil in A/A genotype ovarian cancer patients through clinical trials, with the goal of improving their prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in the study, sign informed consent forms, and have good compliance.
2. After platinum based chemotherapy at Zhejiang Provincial People's Hospital, the efficacy evaluation showed that ovarian cancer patients who achieved disease stability (SD) or disease progression (PD) twice were treated with Fasudil in combination with the original chemotherapy regimen, and were confirmed to have the A/A genotype through genetic testing.

Exclusion Criteria:

* 1.Accompanied by hypotension 2. Bleeding like cerebral hemorrhage 3. Patients with abnormal liver function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  Overall objective tumor response rate

SECONDARY OUTCOMES:
PFS | 3 years
  Progression free Survial

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, M.D., Study Director — Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohta T, Takahashi T, Shibuya T, Amita M, Henmi N, Takahashi K, Kurachi H. Inhibition of the Rho/ROCK pathway enhances the efficacy of cisplatin through the blockage of hypoxia-inducible factor-1alpha in human ovarian cancer cells. Cancer Biol Ther. 2012 Jan 1;13(1):25-33. doi: 10.4161/cbt.13.1.18440. PMID 22336585
- [Background] Wei L, Surma M, Shi S, Lambert-Cheatham N, Shi J. Novel Insights into the Roles of Rho Kinase in Cancer. Arch Immunol Ther Exp (Warsz). 2016 Aug;64(4):259-78. doi: 10.1007/s00005-015-0382-6. Epub 2016 Jan 2. PMID 26725045
- [Background] McLeod R, Kumar R, Papadatos-Pastos D, Mateo J, Brown JS, Garces AHI, Ruddle R, Decordova S, Jueliger S, Ferraldeschi R, Maiques O, Sanz-Moreno V, Jones P, Traub S, Halbert G, Mellor S, Swales KE, Raynaud FI, Garrett MD, Banerji U. First-in-Human Study of AT13148, a Dual ROCK-AKT Inhibitor in Patients with Solid Tumors. Clin Cancer Res. 2020 Sep 15;26(18):4777-4784. doi: 10.1158/1078-0432.CCR-20-0700. Epub 2020 Jul 2. PMID 32616501
- [Background] Ogata S, Morishige K, Sawada K, Hashimoto K, Mabuchi S, Kawase C, Ooyagi C, Sakata M, Kimura T. Fasudil inhibits lysophosphatidic acid-induced invasiveness of human ovarian cancer cells. Int J Gynecol Cancer. 2009 Dec;19(9):1473-80. doi: 10.1111/IGC.0b013e3181c03909. PMID 19955921